CLINICAL TRIAL: NCT02184702
Title: Effects of Shoulder Edema on Intubated Tube in Patients Undergoing Shoulder Arthroscopy
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Collaborators: Fresenius Kabi Korea (Unknown)
Responsible Party: Principal Investigator, Sira Bang, Assistant professor, Inje University
Other Study IDs: IIT-2014-192
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Arthroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- shoulder arthroscopy

SUMMARY:
Intubation is needed in general anesthesia and appropriate cuff pressure is important to avoid trauma or postoperative sore throat and aspiration. Shoulder arthroscope uses some amount of irrigation fluid and it can influence to cuff pressure. Therefore, we will measure cuff pressure during shoulder arthroscope.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1,2 Age 20-65

Exclusion Criteria:

* emergency operation anticipated difficult intubation chronic obstructive lung disease recent upper respiratory infection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patints who undergoing shoulder arthroscopy American Society of Anesthesiologists (ASA) 1,2
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Direct intracuff pressure measurement technique using manometer | every one hour during operarion

CONTACTS AND LOCATIONS:
Overall Officials: Sira Bang, MD, PhD, Principal Investigator — Inje University Seoul Paik Hospital, Seoul, Korea
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, Korea, Seoul, Jung-Gu, South Korea